CLINICAL TRIAL: NCT00546650
Title: A Phase I, Single Center, Open Label, Randomized, Single-Dose, Five-Way Crossover Study to Compare the Pharmacokinetics of NP101 (Sumatriptan Iontophoretic Transdermal Patch) With Three Formulations of Imitrex® in Healthy Volunteers
Brief Title: Phase I Study to Compare NP101(Sumatriptan Iontophoretic Transdermal Patch) With Three Formulations of Imitrex®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP101-005
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Focus of study is to compare pharmacokinetics
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): NP101 patch applied to the upper arm and left in place for 4 hours. The NP101 patch is designed to deliver ~ 10 mg of sumatriptan utilizing up to 600 mA minutes.
  Interventions: Drug: Sumatriptan succinate
- B (Active Comparator): Sumatriptan succinate (Imitrex®) tablet: 100 mg orally.
  Interventions: Drug: Sumatriptan succinate
- C (Active Comparator): Sumatriptan succinate (Imitrex®) injection: 6 mg subcutaneously (SQ).
  Interventions: Drug: Sumatriptan succinate
- D (Active Comparator): Sumatriptan (Imitrex®) nasal spray: 20 mg (one spray) intranasal (IN) into one nostril.
  Interventions: Drug: Sumatriptan succinate
- E (Experimental): NP101 patch applied to the upper arm and left in place for 4 hours. The NP101 patch is designed to deliver ~ 10 mg of sumatriptan utilizing up to 600 mA minutes.
  Interventions: Drug: Sumatriptan succinate

INTERVENTIONS:
Drug: Sumatriptan succinate — NP101 iontophoretic transdermal system
  Arms: A; E
Drug: Sumatriptan succinate — oral, subcutaneous, and intranasal formulations
  Arms: B; C; D

SUMMARY:
The primary objective is to compare the pharmacokinetics (PK) of NP101 with the currently approved oral, injection and nasal spray formulations of Imitrex® in healthy volunteers and to assess the bioavailability relative to the 6 mg subcutaneous injection.

The secondary objective is to evaluate the safety of NP101 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 65 years.
* Women of childbearing potential must be using a medically acceptable form of birth control for the duration of the study, and must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1 for all periods.
* Subjects must have body mass index (BMI) of 18 to 30 kg/m2 inclusive.
* Subjects must be able to communicate effectively with the study personnel.
* Subjects must have, in the investigator's opinion, no clinically significant disease or abnormal laboratory values as determined by medical and psychiatric history, physical examination, or laboratory evaluations conducted at the screening visit or on clinic admission.
* Subjects must have a 12-lead ECG without any clinically significant abnormalities of rate, rhythm, intervals or conduction, as determined by the investigator.
* Subjects must be nonsmokers, defined as having not used any tobacco products in the 6 months before screening.
* Subjects must have not consumed alcoholic beverages, poppy seeds, grapefruit, and/or grapefruit juice within 72 hours prior to admission to the clinic for Period 1 and for the duration of the study.
* Subjects must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.
* The subject must be likely to complete the entire study.

Exclusion Criteria:

* Female subjects who are pregnant or breast feeding or planning a pregnancy during the study.
* A known hypersensitivity to sumatriptan or other triptan agents or the recipients of any of the formulations.
* Subject currently has hypertension with blood pressure outside of normal range for age group.
* Subject has hemiplegic or basilar migraine.
* Subject has severe hepatic impairment.
* Subject has any skin irritation or disease that might interfere with absorption of study drug or skin irritation assessment, including eczema, psoriasis, melanoma, or acne.
* Subject has a tattoo that might interfere with skin erythema examination.
* Subject has a positive test result for hepatitis B, or C or is known to be HIV positive or have a medical history of AIDS.
* Subject who has been administered an injectable drug, except for local anesthetic or birth control, within 30 days prior to the initial study drug administration.
* Subject who requires any medication on a regular basis.
* Subject with a history of malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Subject with a hemoglobin (Hgb) level of less than 7.5 mmol/L.
* Subject has a history, symptoms, or signs of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes.
* Recent (within one year of screening) history of alcohol abuse, illicit drug use, physical dependence to any opioid, or recent (within one year of screening) history of drug abuse or addiction.
* Concurrent use of prescription (Rx) or over-the-counter (OTC) medications or natural medicine (herbal) products.
* Subject is currently taking MAO-A inhibitors
* Receipt of an investigational drug or participation in any clinical study within 90 days prior to study entry.
* Donation of blood or blood products within 8 weeks prior to study entry.
* Positive urine drug screen, including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates.
* Subject who is considered by the investigator or NuPathe, for any reason, to be an unsuitable candidate for receiving sumatriptan, or as being unsuitable for any other reason as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Blood samples to be drawn at pre-dose (within 15 minutes prior to dosing) and at 0.25, 0.50, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 16 hrs post dose.
  The primary objective was to compare the pharmacokinetics (PK) of NP101 (sumatriptan iontophoretic transdermal patch) with the currently approved oral, subcutaneous injection and nasal spray formulations of Imitrex® in healthy volunteers and to assess the bioavailability relative to the 6 mg subcutaneous injection.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States